CLINICAL TRIAL: NCT04154774
Title: A Single-Dose, Open-Label Study to Evaluate the Pharmacokinetics of Apalutamide in Subjects With Severe Hepatic Impairment Compared With Subjects With Normal Hepatic Function
Brief Title: A Study of Apalutamide in Participants With Severe Hepatic Impairment Compared With Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108714; 56021927PCR1026 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Participants with Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment will receive single oral dose of apalutamide on Day 1 under fasted condition.
  Interventions: Drug: Apalutamide
- Group 2: Participants with Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive single oral dose of apalutamide on Day 1 under fasted condition.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Apalutamide will be administered orally.
  Other Names: JNJ-56021927

SUMMARY:
The purpose of this study is to characterize the single-dose pharmacokinetic (PK) of apalutamide in participants with severe hepatic impairment relative to participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Participants must not have hepatic encephalopathy greater than or equal to (>=) Grade 3 (for participants with severe hepatic impairment) where the participant lacks the capacity to provide informed consent as judged by the investigator. Mild or moderate hepatic encephalopathy that would not impede informed consent in the investigator's judgment is permitted
* Participants with normal hepatic function must be in good health with no clinically significant findings from medical history, physical examination, vital signs, and laboratory evaluation, unless deemed not clinically significant by the investigator
* Participants with normal hepatic function must have serum creatinine within normal limits and Creatinine Clearance (CrCL) greater than (>) 60 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) as calculated per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation
* Participants with severe hepatic impairment must have a total Child-Pugh score of 10 to 15 inclusive, as determined by the investigator during screening and on Day -1 prior to study drug administration. Source documents to substantiate the clinical diagnosis (for example, ultrasonography, liver biopsy, liver/spleen scan, laboratory results or clinical findings), and medical history will be reviewed and signed by the investigator
* Participants with severe hepatic impairment must have CrCL >= 45 mL/min/1.73 m^2 as calculated per CKD-EPI Creatinine Equation

Exclusion Criteria:

* Use of thyroid hormone replacement therapy
* Participants with normal hepatic function with presence of sexual dysfunction (abnormal libido, erectile dysfunction, etc.) or any medical condition that would affect sexual function
* Participants with normal hepatic function who have Hepatitis A immunoglobulin M positivity, Hepatitis B surface antigen (HBsAg) positivity, positive serology for Hepatitis B or Hepatitis C antibodies. Hepatitis B surface antibody positivity is not exclusionary if participant can provide evidence of Hepatitis B vaccination
* Participants with severe hepatic impairment who have acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment in the judgment of either the investigator or the sponsor's medical monitor
* Participants with severe hepatic impairment previously diagnosed with hepatocellular carcinoma

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Area Under Concentration-time Curve from Time 0 to Infinite Time (AUC[0-infinity]) of Apalutamide | Up to Day 57
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C (last)/ lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to the time of the last measurable concentration, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under Concentration-time Curve from Time 0 to the Time of the Last Concentration (AUC[0-last]) of Apalutamide | Up to Day 57
  AUC(0-last) is defined as the time 0 to the time of the last measurable (non-below quantification limit) concentration of apalutamide calculated by linear-linear trapezoidal summation.
Peak Plasma Concentration (Cmax) of Apalutamide | Up to Day 57
  Cmax is defined as peak observed plasma concentration of the drug.

SECONDARY OUTCOMES:
Number of Participants with Adverse Event as a Measure of Safety and Tolerability | Up to 78 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Homestead Associates in Research Inc, Homestead, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, Tampa, Florida
  - VGR & NOCCR - Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency